CLINICAL TRIAL: NCT04537741
Title: Coronary CT Angiography in Non ST-elevation Myocardial Infarction (NSTEMI) - a Way to Reduce Unnecessary Invasive Investigations
Brief Title: Coronary CT Angiography in Non ST-elevation Myocardial Infarction
Acronym: CT-NSTEMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Helse Nord-Trøndelag HF (Other); Namsos Hospital (Other); Volda Hospital (Other); Kristiansund Hospital (Other); Molde Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 45965
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Non-ST Elevated Myocardial Infarction
Keywords: Coronary angiography; Angiography, CT; NSTEMI; CCTA; CT-FFR
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Single arm study where all patients being included will undergo CCTA before invasive coronary angiography
Masking Description: CCTA will be analysed at a core lab with no information of the results from invasive angiography or whether coronary revascularization was performed or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSTEMI scheduled for angiography (Experimental)
  Interventions: Procedure: Coronary CT angiography; Procedure: Invasive coronary angiography

INTERVENTIONS:
Procedure: Coronary CT angiography — all patients being included will undergo CCTA before invasive coronary angiography
Procedure: Invasive coronary angiography — all patients being included will undergo CCTA before invasive coronary angiography

SUMMARY:
Non ST-elevation myocardial infarction (NSTEMI) represents 70-75% of all myocardial infarctions. Current guidelines recommend invasive angiography and this patient group represents a major burden on the invasive catheterization laboratories and the health care system.

The coronary pathology found in NSTEMI-patients varies substantially, ranging from structurally normal vessels, non-obstructive atherosclerosis to severe multivessel disease. 30-40 % of patients with NSTEMI undergoing invasive coronary angiography do not undergo revascularization. If these patients could be identified by a non-invasive method like coronary CT angiography (CCTA), an invasive procedure with the potential risk for complications could be avoided. Furthermore, less patients would need transfer to an invasive center. Both for patients and for health care costs this would be of major benefit.

The quality of CCTA images has improved during the years, and radiation dose has decreased. Due to technological development it is now possible to perform high quality coronary CCTA with a very low radiation dose (1-1.5 mSv) compared to a radiation dose of 3-4 mSv for invasive coronary angiography.

The overall aim of the project is to define a subpopulation of NSTEMI patients that preferably should undergo CCTA as the first step in imaging of the coronary arteries and thus potentially be saved from an unnecessary invasive investigation. This would result in less patient discomfort, less patient risk and reduced health care costs. Patients with a clinical indication for invasive angiography according to current guidelines will undergo CCTA prior to the invasive investigation. The ability of CCTA to identify those with no need for revascularization will be assessed using invasive angiography as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* admitted to a local hospital with NSTEMI type 1 or type 2 based on clinical criteria
* indication for invasive coronary angiography according to current guidelines

Exclusion Criteria:

* indication for immediate (< 2 hours) invasive strategy according to guidelines
* GRACE score > 140
* not willing to provide written informed consent
* previous coronary revascularization
* estimated glomerular filtration rate < 30 mL/min/1,73m2
* allergic reactions to contrast agents impeding for safe examinations
* > 2 hypokinetic segments on echocardiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The number of patients with coronary artery disease in need for revascularization as defined by invasive coronary angiography including invasive iFR/FFR | 1 month
  For the primary endpoint analysis will be performed on patient level

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, prof dr md, Study Director — St Olavs Hospital, Clinic of Cardiology; Øystein Risa, Study Director — Norwegian University of Science and Technology, ISB
Locations (8):
- Norway (8):
  - Ålesund Hospital, Cardiac Unit, Ålesund
  - Kristiansund Hospital, Cardiac Unit, Kristiansund
  - Levanger Hospital, Cardiac Unit, Levanger
  - Molde Hospital, Cardiac Unit, Molde
  - Namsos Hospital, Cardiac Unit, Namsos
  - Orkdal Hospital, Cardiac Unit, Orkdal
  - St Olavs Hospital Clinic of Cardiology, Trondheim
  - Volda Hospital, Cardiac Unit, Volda

IPD SHARING:
Plan to Share IPD: No